CLINICAL TRIAL: NCT07186686
Title: Development of the AMENUCED Program and Evaluation of Its Feasibility in Adults With Type 2 Diabetes: A Pre-Post Study
Brief Title: Feasibility Study of AMENUCED Program in Type 2 Diabetes
Acronym: AMENUCED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Full-time professor, Universidad de Sonora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMENUCED-DT2-01
Record Dates: First submitted 2025-09-02; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Diabete Type 2
Keywords: Type 2 Diabetes Mellitus; Pilot Study; Feasibility; Self management education; Lifestyle intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMENUCED Intervention Group (Experimental): Participants will receive the AMENUCED program including medical care, nutritional counseling, and structured sessions focused on behavioral change and diabetes education. The study is designed to assess the feasibility and acceptability of the AMANUCED program in adults with Type 2 Diabetes. This intervention does not involve any pharmacological or device-based components.
  Interventions: Other: Participants will receive the AMENUCED program including medical care, nutritional counseling, and structured sessions focused on behavioral change and diabetes education.

INTERVENTIONS:
Other: Participants will receive the AMENUCED program including medical care, nutritional counseling, and structured sessions focused on behavioral change and diabetes education. — Medical Attention: Medical management will be provided by a physician who will assess the participant at the beginning and end of the intervention. The physician will be responsible for pharmacological treatment and follow-up throughout the process.
  Nutritional Attention: Nutritional consultations will be provided by a registered nutritionist over a three-month period, with sessions held weekly. During each consultation, the participant will receive an individualized nutrition plan based on scientific evidence and dietary recommendations. The plan will be tailored to the participant's specific needs, including metabolic control and a hypocaloric intake (ranging from 1200 to 1800 kcal), with the goal of achieving a 5-10% reduction in body weight.
  Behavioral Lifestyle Change Program: The behavior modification program used in the Action for Health in Diabetes Program (Look AHEAD) study will be adapted to include diabetes self-management activities through a structured manual.

SUMMARY:
Type 2 diabetes is characterized by progressive resistance to the effects of insulin, along with deficient insulin production. In Mexico, it affects 18.4% of adults and is the second leading cause of death. According to ENSANUT 2023, 74.2% of adults with diabetes have poor glycemic control. Achieving adequate glycemic control requires multiple interventions. The AMENUCED program is multicomponent and includes medical care, nutritional guidance, lifestyle support, and diabetes education. Each component has independently shown positive outcomes in diabetes management, yet few Mexicans receive this comprehensive care.

This study aims to develop the AMENUCED program and evaluate its feasibility (acceptance and retention) after a 3-month intervention in adults with type 2 diabetes.

A pre-post pilot study will be conducted. The primary outcome is program feasibility, while secondary outcomes include HbA1c, body weight, BMI, waist circumference, body fat, fasting glucose, plasma lipids, blood pressure, mental health aspects, and diabetes knowledge. Statistical analysis will be exploratory, using paired t-tests or Wilcoxon tests to compare pre- and post-intervention data, and McNemar's test to compare proportions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 and ≤65 years
* Residing in Hermosillo, Sonora
* Body Mass Index (BMI) ≥25
* Prior diagnosis of Type 2 Diabetes
* Individuals who cannot read or write may be included if accompanied by someone willing to attend sessions and assist with comprehension
* Must have active medical insurance

Exclusion Criteria:

* Diabetes-related complications, including:

  * Advanced diabetic nephropathy
  * Neuropathy
  * Retinopathy
  * Cardiovascular or cerebrovascular diseases
* History of severe hypoglycemia
* Significant metabolic dysregulation (HbA1c ≥10%)
* Use of insulin, sulfonylureas, or meglitinides
* Pregnancy or breastfeeding within the past 6 months
* Diagnosed psychiatric disorders
* Consumption of ≥14 alcoholic beverages per week
* Serious illnesses (e.g., cancer, liver failure, kidney disease)
* Chronic use of corticosteroids
* Plans to relocate during the study period
* Weight loss greater than 5% in the past three months
* History of bariatric surgery
* Any other medical, psychiatric, or behavioral condition that, in the investigator's judgment, may interfere with participation in the intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the AMENUCED Program | Baseline to 12 weeks post intervention
  Acceptance will be assessed by participant ratings using a 1-10 scale (where 1= lowest acceptance and 10 = highest acceptance) for each component of the program, including educational content, delivery format, and perceived usefulness. Unit of measure: Score 1 - 10.
Retention in the AMENUCED Program | Baseline to 12 weeks post intervention.
  Retention will be measured by the percentage of participants who remain in the program. Unit of Measure: Percentage of participants (%)

SECONDARY OUTCOMES:
Change in Glycated Hemoglobin | Baseline and 12 weeks post-intervention
  Measured using standardized blood tests to assess glycemic control. Unit of Measure: %
Change in body fat | Baseline and 12 weeks post-intervention
  Measured in using medical body composition analyzer (Seca mBCA 514) under standardized conditions. Unit of measure (kg of body fat)
Change in Body Mass Index | Baseline and 12 weeks post-intervention
  Calculated as weight (kg) divided by height squared (m²), using standardized equipment and protocol. Unit of measure: kg/m²
Change in waist circumference | Baseline and 12 weeks post-intervention
  Measured with anthropometric tape (Lufkin Executive W606PMMX) at the umbilical level. Unit of measure: cm
Change in Blood Pressure | Baseline and 12 weeks post-intervention
  Systolic and diastolic blood pressure will be measured using an Omron digital sphygmomanometer (HEM-907XL) on the upper arm, following American Heart Association guidelines. Unit of Measure: mmHg
Change in Health-Related Quality of Life | Baseline and 12 weeks post-intervention
  Assessed using the "SF-36 Health Survey", with scores ranging from 0 = worst possible health status, to 100 = best possible health status. Unit of measure: 0 - 100
Change in Fasting Glucose | Baseline and 12 weeks post-intervention
  Measured via standardized laboratory testing. Unit of Measure: mg/dL
Change in Perceived Stress | Baseline and 12 weeks post-intervention.
  Assessed using "The Coping Stress Questionnaire (CAE): Validation in a Mexican Sample". The CAE includes seven subscales: problem-solving focus, negative self-focus, positive reappraisal, open emotional expression, avoidance, social support seeking and religious coping. Participants rate each item on a 6-point Likert scale (0 = never, 5 = always). Higher scores indicate more frequent use of the corresponding coping strategy. Use of Measure: Subscale scores (range: 0-5 per item; total score varies by subscale)
Change in Depression Symptoms | Baseline and 12 weeks post intervention.
  Assessed using the Beck Depression Inventory-II, a 21 item self-report questionnaire designed to measure the severity of depression. Each item is rated on a 4 point Likert scale (0 = not al all, 3 = severe), with total scores ranging from 0 to 63. Higher scores indicate greater severity of depressive symptoms. Unit of Measure: Total score range 0 - 63
Change in Anxiety Symptoms | Baseline and 12 weeks post intervention.
  Assessed using the "Beck Anxiety Inventory (BIA), a 21 item self report questionnaire designed to measure the severity of anxiety in adults. Each item is rated on a 4 point likert scale (0 = not al all, 3 = severely), with total scores ranging from 0 to 63. Higher scores indicate greater severity of anxiety symptoms. The BAI has demonstrated strong psychometric properties in general Mexican populations. Unit of Measure: Total score range 0 - 63
Change in Diabetes Knowledge | Baseline and 12 weeks post intervention.
  Assessed using the "24 - item version of the Diabetes Knowledge Questionnaire (DKQ-24), developed and validated in Spanish for Mexican-American populations. Each item is scored as correct or incorrect, with total scores ranging from 0 to 24. Higher scores indicate greater diabetes-related knowledge. Unit of Measure: Total score, range 0 - 24
Change in Total Cholesterol | Baseline and 12 weeks post intervention
  Measured via standardized laboratory testing. Unit of Measure: mg/dL
Change in HDL Cholesterol | Baseline and 12 weeks post intervention
  Measured via standardized laboratory testing. Higher values indicated better cardiovascular profile. Unit of Measure: mg/dL
Change in LDL Cholesterol | Baseline and 12 weeks post intervention
  Measured via standardized laboratory testing. Unit of Measure: mg/dL
Change in Triglycerides | Baseline and 12 weeks post intervention
  Measured via standardized laboratory testing. Unit of Measure: mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora 83000, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared, as this study corresponds to a pilot phase with a small sample size.